CLINICAL TRIAL: NCT05343910
Title: The Effect of Aroma Massage on Constipation in Elderly
Brief Title: The Effect of Aroma Massage on Constipation
Acronym: aromatherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Didem Lafci, Principal Investigator, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MersinUniversty
Record Dates: First submitted 2022-03-23; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Constipation
Keywords: aroma massage; constipation; elderly; nursing
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aromatherapy massage group (Experimental): Experimental: aromatherapy massage group The oil mixture used in this study (1:, 1:, 1: 1, 20cc rosemary, 20cc mint, 20cc ginger, 20cc black pepper), 80% of the mixture obtained from the total 4% (3.2cc) carrier oil (100% almond oil=96.8cc) and then combined with abdominal massage. Before implementing the procedure in the experimental group (n=25), information about what an abdominal and aroma massage is, how long it will take, and how it will be applied was provided to the participants. The older adult participants in the experimental group were applied aroma massage through gentle movements with slight pressure for 15 min a day, five days a week for three weeks.
  Interventions: Other: Aroma massage
- Control group (No Intervention): Individuals in the control group (n=24) did not receive any type of aroma massage application.

INTERVENTIONS:
Other: Aroma massage — The older adult participants in the experimental group were applied aroma massage through gentle movements with slight pressure for 15 min a day, five days a week for three weeks.
  Arms: Aromatherapy massage group

SUMMARY:
Advancing age arising changes in health status and systems adversely affect the quality of life of the elderly and the elderly face many complex health problems. Constipation is one of the common problems in the elderly. Therefore, The aim of this study is to examine effects of aromatherapy massage on constipation in the elderly.

DETAILED DESCRIPTION:
Old age is a physiological period of life in which various changes take place, meaning that the elderly must be given special consideration as a group with regard to health care. Advancing age arising changes in health status and systems adversely affect the quality of life of the elderly and the elderly face many complex health problems. Constipation is one of the common problems in the elderly. Insufficient liquid intake, insufficient or unsuitable diet, decreased mobility, the side effects of medication, underlying diseases, and rectal sensory-motor dysfunction are among the causes of constipation in the elderly. Constipation is a preventable and treatable problem, which if left untreated can cause physical and associated psychological problems such as back and waist pain, rectal pressure, loss of appetite, confusion, incontinence, nausea and vomiting, urinary dysfunction, fissure, rectal prolapse, hemorrhoids, intestinal obstruction, and syncope. Constipation can be managed using pharmacological methods, such as laxatives, enemas, suppositories, along with nonpharmacological procedures, such as changes in nutritional habits, fluid intake, education, activities to develop healthy intestinal habits, exercise, massage, aroma massage, biofeedback, stress management and acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older
* Communication and cooperation can be established
* Conscious,, agreeing to participate in the research,
* Decreasing bowel movements, not able to deactivate for 3 days or more
* Living more than two of the complaints related to defecation, who have not undergone intestinal surgery before
* Lesion or infection that disrupts skin integrity in the abdominal region, elderly without any problems such as heart disease and dementia

Exclusion Criteria:

* had language problems
* were below 65 years of age and
* refused to participate in the study.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2013-03-01 (Actual); Study Completion 2013-03-01 (Actual)

PRIMARY OUTCOMES:
Stool consistency | change from before intervention, 3rd and 4th week of intervention
  Small as marble, hard (1 point) Bulky, hard (2 points) Normal (3 points) Soft (4 points) Juicy (5 points)
  7-day total value for stool consistency / 7-day total number of stools
Amount of stool | change from before intervention, 3rd and 4th week of intervention
  None (0 points) Less than the previous stool (1 point) Normal (2 points) a lot (3 points) 7-day total value for stool amount / 7-day total number of stools
Straining during defecation | change from before intervention, 3rd and 4th week of intervention
  Defecation without straining (1 point) Straining at the beginning of defecation (2 points) Straining at half defecation (3 points) Straining during the entire defecation (4 points)
  Obtained 7 days for straining during defecation total value / total number of defecations in 7 days
38 / 5.000 Çeviri sonuçları Full after defecation feeling of inability to ejaculate | change from before intervention, 3rd and 4th week of intervention
  None after defecation (0 points) Present after defecation (1 point)
  7 for the feeling of incomplete ejaculation after defecation. total value obtained per day / total number of defecations in 7 days
Number of defecations | change from before intervention, 3rd and 4th week of intervention
  How many defecations per day
  Total number of defecations in 7 days / 7

CONTACTS AND LOCATIONS:
Overall Officials: Mağfiret Kaşıkçı, Prof., Study Director — Ataturk University
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No